CLINICAL TRIAL: NCT00938730
Title: A Phase 2, Double-Blind, Double-Dummy, Randomized, Parallel Group Dose Finding Study To Investigate the Safety and Tolerability of YM150 in Subjects With Non-Valvular Atrial Fibrillation and to Compare the Safety and Tolerability With Warfarin
Brief Title: A Study Evaluating Safety and Tolerability of YM150 Compared to Warfarin in Subjects With Atrial Fibrillation
Acronym: OPAL-2
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Astellas Pharma Inc (Industry)
Responsible Party: Disclosure Office Europe, Astellas Pharma Europe BV
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: 150-CL-021; 2007-001150-87 (EudraCT Number)
Record Dates: First submitted 2009-07-01; First posted 2009-07-14 (Estimated); Last update posted 2011-01-20 (Estimated); Status verified 2011-01

CONDITIONS: Atrial Fibrillation
Keywords: Nonvalvular Atrial Fibrillation (NVAF); Factor Xa Inhibitor; Stroke; Thromboembolism; Transient Ischemic attack; Anticoagulants; Prevention; YM150; Warfarin
MeSH Terms: conditions — Atrial Fibrillation; Stroke; Thromboembolism; Ischemic Attack, Transient | interventions — Warfarin

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (7):
- 1. YM150, Dose W, twice daily (Experimental)
  Interventions: Drug: YM150
- 2. YM150, Dose X, once daily (Experimental)
  Interventions: Drug: YM150
- 3. YM150, Dose X, twice daily (Experimental)
  Interventions: Drug: YM150
- 4. YM150, Dose Y once daily (Experimental)
  Interventions: Drug: YM150
- 5. YM150, Dose Y twice daily (Experimental)
  Interventions: Drug: YM150
- 6. YM150, Dose Z, once daily (Experimental)
  Interventions: Drug: YM150
- 7. Warfarin (Active Comparator)
  Interventions: Drug: Warfarin

INTERVENTIONS:
Drug: YM150 — oral
  Arms: 1. YM150, Dose W, twice daily; 2. YM150, Dose X, once daily; 3. YM150, Dose X, twice daily; 4. YM150, Dose Y once daily; 5. YM150, Dose Y twice daily; 6. YM150, Dose Z, once daily
Drug: Warfarin — oral
  Arms: 7. Warfarin

SUMMARY:
The purpose of this study is to investigate the optimal daily dose and dose regimen of YM150 in subjects with non-valvular atrial fibrillation (NVAF), primarily based on safety and tolerability data.

ELIGIBILITY:
Inclusion Criteria:

* Subject with paroxysmal, permanent or persistent Nonvalvular Atrial Fibrillation (NVAF)
* Subject has prothrombin time international normalized ratio (INR) of 2.0 or below at the baseline visit

Exclusion Criteria:

* Subject has current or recent (within 12 months prior to screening) history of stroke and/or systemic embolism (including TIA)
* Subject has active bleeding or any condition associated with increased risk of bleeding
* Subject has NVAF secondary to other reversible disorders (e.g. thyrotoxicosis)
* Subject has an indication for warfarin other than AF (including planned cardioversion)
* Subject has had a diagnosis of Acute Coronary Syndrome (ACS), coronary artery bypass graft (CABG) or percutaneous transluminal coronary angioplasty (PTCA) within previous 3 months of screening
* Subject has a diagnosis of left ventricular aneurysm or atrial myxoma
* Subject requires use of prohibited previous and concomitant medication (i.e., thrombolytics [such as tissue Plasminogen Activator (tPA), streptokinase], antiplatelet agents [such as cilostazol, clopidogrel, ticlopidine, dipyridamole], anticoagulants [such as vitamin K antagonists, heparin, unfractionated or low molecular weight heparin, fondaparinux, thrombin inhibitors] and chronic use of nonsteroidal anti-inflammatory drugs [NSAIDs] or acetylsalicylic acid use of >100 mg/day). (see Section 5.1.3 and Appendix 1 for details)
* Subject has active infective endocarditis
* Subject is planned for invasive procedures with potential for bleeding
* Subject has participated in another clinical trial of an investigational drug (including placebo) or device within 30 days (or the limit set by national law, whichever is longer) of signing informed consent for the present study
* Subject has participated in any YM150 clinical trials

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1280 (Actual)
Dates: Start 2009-06; Primary Completion 2010-09 (Actual); Study Completion 2010-09 (Actual)

PRIMARY OUTCOMES:
Incidence of major and clinically relevant non-major bleeding events | Double-blind treatment period (variable, up to 16 months)

SECONDARY OUTCOMES:
Composite and individual incidences of ischemic strokes, TIAs, systemic thrombolic events, ACS, all deaths | Double-blind treatment period (variable, up to 16 months)
Incidence of bleeding events | Double-blind treatment period (variable, up to 16 months)
Assessment of other safety variables | Double blind treatment period (variable, up to 16 months)
Assessment of PK/PD variables | Double-blind treatment period (up to week 12)
Patient Reported Outcomes | Double-blind treatment period (up to week 24)

CONTACTS AND LOCATIONS:
Overall Officials: Use Central Contact, Study Chair — Astellas Pharma Europe B.V.
Locations (140):
- Australia (4):
  - Auchenflower
  - Caboolture
  - Kippa-Ring
  - Victoria
- Vienna, Austria
- Bulgaria (3):
  - Dimitrovgrad
  - Pleven
  - Sofia
- Czechia (5):
  - Besenov
  - Havirov-mesto
  - Prague
  - Tábor
  - Ústí nad Labem
- Estonia (3):
  - Narva
  - Tallinn
  - Tartu
- Paris, France
- Germany (9):
  - Bad Nauheim
  - Berlin
  - Darmstadt
  - Dresden
  - Hagen
  - Kassel
  - Mainz
  - Mannheim
  - Markkleeberg
- Hungary (6):
  - Balatonfüred
  - Budapest
  - Debrecen
  - Mosonmagyaróvár
  - Nyíregyháza
  - Székesfehérvár
- India (9):
  - Ahmedabad
  - Bangalore
  - Hyderabaad
  - Kolkata
  - Madurai
  - Nagpur
  - Nashik
  - Nellore
  - Pune
- Israel (3):
  - Nahariya
  - Nazareth
  - Rehovot
- Japan (26):
  - Asahikawa
  - Atsugi
  - Bunkyō City
  - Daitō
  - Fujisawa
  - Funabashi
  - Hachiōji
  - Higashiibaraki-gun
  - Hiroshima
  - Kanazawa
  - Kasaoka
  - Kishiwada
  - Kitamoto
  - Kiyose
  - Kobe
  - Meguro-ku
  - Morioka
  - Nankoku
  - Sapporo
  - Sendai
  - Shimajiri-gun
  - Shinjyuku-ku
  - Shizuoka
  - Toyama
  - Wako
  - Yokohama
- Malaysia (2):
  - Kuala Lumpur
  - Selangor Darul Ehsan
- Netherlands (3):
  - AD Delft
  - AE Roosendaal
  - BC Amsterdam
- Iloilo City, Philippines
- Poland (10):
  - Bytom
  - Gdynia
  - Katowice
  - Kielce
  - Krakow
  - Lodz
  - Lublin
  - Torun
  - Warsaw
  - Wroclaw
- Russia (11):
  - Arkhangelsk
  - Chelyabinsk
  - Moscow
  - Novosibirsk
  - Omsk
  - Saint Petersburg
  - Saratov
  - Smolensk
  - Tomsk
  - Tula
  - Tyumen
- Slovakia (6):
  - Bardejov
  - Dolný Kubín
  - Komárno
  - Košice
  - Liptovský Hrádok
  - Martin
- South Africa (9):
  - Bellville
  - Benoni
  - Centurion
  - Chatsworth
  - Moreletapark
  - Somerset West
  - Tongaat
  - Umhlanga
  - Worcester
- South Korea (4):
  - Busan
  - Gwangju
  - Incheon
  - Seoul
- Spain (3):
  - Murcia
  - Seville
  - Viladecans
- Thailand (2):
  - Bangkok
  - Chiang Mai
- Ukraine (11):
  - Cherkassy
  - Donetsk
  - Ivano-Frankivsk
  - Kharkiv
  - Kyiv
  - Lutsk
  - Lviv
  - Odesa
  - Ternopil
  - Vinnytsia
  - Zaporizhzhya
- United Kingdom (8):
  - Addlestone
  - Bath
  - Birmingham
  - Dundee
  - East Horsley
  - London
  - Soham
  - Southampton